CLINICAL TRIAL: NCT05738044
Title: Multi-omics Analyses of Airway Host-microbiome Interaction in Chronic Obstructive Pulmonary Disease and Bronchiectasis Identify Potential Therapeutic Interventions
Brief Title: Multi-omics Studies of Host-microbiome Interaction in Chronic Obstructive Pulmonary Disease and Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COPD-BE
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: COPD Exacerbation; Bronchiectasis With Acute Exacerbation
Keywords: Chronic Obstructive Pulmonary Disease; Bronchiectasis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients: Patient meets diagnose of COPD refering to "Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2022" will be included.
  Interventions: Other: No intervention
- Bronchiectasis patients: Patients diagnosed with bronchiectasis (according to the Chinese consensus, patient's previous chest CT examination must show bronchiectasis)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Chronic obstructive pulmonary disease (COPD) and bronchiectasis are common chronic respiratory diseases in China. COPD is characterized by irreversible lung function decline due to airway inflammation, emphysema and alveolar destruction. Bronchiectasis is characterized by permanent bronchiectasis, its main clinical symptoms are cough, dyspnea, hemoptysis and recurrent respiratory tract infections. The incidence and prevalence of bronchiectasis have assumed continuously grows in global. Airway microbiota, whose alterations play an important role in the occurrence and development of bronchiectasis, form a complex ecosystem interacted with host cells and various biotic and abiotic factors in the microenvironment. Additionally, mounting evidence suggests that the airway microbiome is associated with COPD phenotypes and endotypes, and that dysbiosis contributes to airway inflammation. However, the mechanisms remain poorly understood, owing to limited knowledge of microbial functional properties, metabolic activities and cross-talk with the host immune system. The investigators aim to collect sputum specimen and perform multi-omic analysis on patients with COPD and bronchiectasis in seven clinical centres in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bronchiectasis (according to the Chinese consensus, patient's previous chest CT examination must show bronchiectasis) or COPD (according to GOLD 2022).
* Patients with age ≥18 years old.
* Written informed consent.

Exclusion Criteria:

* Pregnancy or lactation, or those without taking effective contraceptive measures
* Subjects with a history of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders
* Subjects with a history of alcohol or illicit drug abuse
* Subjects with any of the following pulmonary diseases: active tuberculosis, pulmonary embolism, pneumothorax, multiple huge bullae, uncontrolled asthma, acute exacerbation of chronic bronchitis or extremely severe COPD
* Diagnosis of chronic gastrointestinal disease, heart disease, diabetes, severe renal insufficiency (GFR < 30ml/min) or immunodeficiency
* Participated in any interventional clinical trial within 3 months before enrolment.
* Poor compliance or inability to cooperate as judged by the doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients enrolled in this study should meet the bronchiectasis diagnositc criteria according to the Chinese consensus or COPD diagnositc criteria according to GOLD 2022.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of lung microbiome in COPD and bronchiectasis patient between exacerbation and clinically stable stage | Day0 and week 10
  The lung microbiome of COPD and bronchiectasis patients will be defined from sputum samples using traditional bacterial culture and 16S rRNA sequencing.

SECONDARY OUTCOMES:
Change of lung metabolomics in COPD and bronchiectasis patient between exacerbation and clinically stable stage | Day0 and week 10
  The lung microbiome of COPD and bronchiectasis patients will be defined from sputum samples using liquid chromatography-mass spectrometry (LC-MS)-based metabolomics approach.
Change of lung proteomics in COPD and bronchiectasis patient between exacerbation and clinically stable stage | Day0 and week 10
  The lung microbiome of COPD and bronchiectasis patients will be defined from sputum samples using Olink multiplex panel.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China